

# Addis Ababa Science and Technology University

CONSENT FORM August 19 2022

This Consent Form is for children who are invited to participate on the study "assessment of nutrient profile, nutritional status, development and severity of children with autistic spectrum disorder in comparison with typically developing children in Addis Ababa, Ethiopia"

| CONTACT AND PROJECT DETAILS | |
|---|---|
| Researcher's Full Name: | Feven Yirgu (MSc candidate) |
| Contact Details: | kirkos sub-city, woreda 04, P.no. 0921029147 |
| Supervisor's Full Name: | Abera Belay (PhD) |
| Project Title: | Assessment of nutrient profile, nutritional status, development and severity of children with autistic spectrum disorder in comparison with typically developing children in Addis Ababa, Ethiopia |

This Informed Consent Form has two parts:

- Information Sheet (to share information about the research)
- Certificate of Consent (for signatures if you agree to take part)

#### **SECTION I: INFORMATION SHEET**

#### Introduction

My name is Feven Yirgu, MSc candidate in Food Science and Nutrition in Addis Ababa Science and Technology University. I am doing my research on Assessment of nutrient profile, nutritional status, development and severity of children with autistic spectrum disorder in comparison with typically developing children in Addis Ababa, Ethiopia. I am going to give you information and invite you to be part of this study.

### **Purpose of the study**

Proper nourishment and a balanced diet is important for every child and children with autistic spectrum disorder (ASD) are especially vulnerable to various form of malnourishments as result of the eating behaviour and various physiological conditions related with the disorder. Given that this area is under researched this study aims to assess the nutritional status of ASD children as compared to their typically developing peers.

## **Type of Research Intervention**

This research will involve height, weight and middle upper arm circumference measurements, urine iodine concentration, three days food diary, childhood rating scale analysis and eating behaviour and food frequency questioner

### **Participant selection**

Inclusion criteria: case

• Children already diagnosed with ASD



# Addis Ababa Science and Technology University

CONSENT FORM August 19 2022

• School aged (4-18) Exclusion criteria: case

• use of special supplements and heavy medication

• critical chronic disease such as cancer, HIV AIDs

Inclusion criteria: control

• Matched school age children

Exclusion criteria: control

- use of special supplements and heavy medication
- critical chronic disease such as cancer, HIV AIDs

#### **Procedures and Protocol**

Anthropometry – measuring weight, height and upper arm circumference using a weight board, height board and flexible measuring tape

Urine sample collection - 60 ml. urine samples is collected from each child by trained Autistic child handlers, at the child's period of urinary stimulation using sample collection cups.

Three day food diary – recording of all foods consumed for a three days period

Proximate analysis - collecting 50gm sample of food in sample collection bags from each meal consumed throughout the day by the researcher and legal guardians for analysis.

Childhood autism rating scale (CARS) – using the CARS rating booklet performed by a medical practitioner to score the children on the questions described

Dietary assessment – collecting food frequency, eating behaviour, dietary diversity using a questioner

**Note:** Please ask if there are some words that you do not understand, will go through the information & take time to explain. If you need to stop your good participation, you are allowed to stop your participation any time.



# Addis Ababa Science and Technology University

CONSENT FORM August 19 2022

#### **SECTION 2: CERTIFICATION**

| Pa | ar | tici | pant | Cer | tifi | cat | io | n |
|----|----|------|------|-----|------|-----|----|---|

In signing this form, I confirm that:

- I have read the Participant Information Sheet and the nature and purpose of the research project has been explained to me.
- I understand the procedure and agree to take part.
- I understand the purpose of the research project and my involvement in it.
- I understand that while information gained during the study may be published, I will not be identified and my personal results will remain confidential, unless required by law.

| Participant Signature | Name | Date |
|-----------------------|------|------|

| Researcher Certification |
|---|
| I have explained the study to subject and consider that he/she understands what is involved. |

Researcher Signature

Name

Date



### Addis Ababa Science and Technology University

**CONSENT FORM** August 19 2022

#### ETHICAL CLEARANCE

Addis Ababa Science and Technology University አዲስ አበባ ማድንስና ቴክኖሎጂ ዩኒቨርሲቲ

# TO WHOM IT MAY CONCERN

The Institutional Ethical Approval Board of Addis Ababa Science and Technology University in its meeting held on 2nd August 2021 has examined the study project of Feven Yirgu (Principal Investigator), entitled "ASSESSMENT OF NUTRIENT PROFILE, NUTRITIONAL STATUS, DEVELOPMENT AND SEVERITY OF CHILDREN WITH AUTISTIC SPECTRUM DISORDER IN COMPARISON WITH TYPICALLY DEVELOPING CHILDREN IN ADDIS ABABA, ETHIOPIA. The proposal was approved for implementation.

Accordingly, our University's Ethical Approval Board has evaluated the researcher's study Propasal as per the University's Research Ethics evaluation criteria and assures that his study has fulfilled all the required criteria on the day of March 17, 2021.

Therefore; our good Office has provide this Ethical Clearance/Approval letter to Feven Yirgu.

Best Regards,

Abraham Debebe Woldeyohannes (PhD) Research and Technology Transfer Vice President



#### CC:

- Research and Technology Transfer Vice President Office
- · Research Directorate
- · Institutional Ethical Approval Board
- · Feven Yirgu.

AASTU

መልስ ሲፅፉ የኛን ቁጥር ይጥቀሱ

251-11-462-40-11

Web site: www.aastu.edu.et

When replying please indicate our reference No. 🖂 16417 አዲስ አበባ አ ትዮጵያ